CLINICAL TRIAL: NCT05528562
Title: PrEP Rapid Access: An Open Pilot Study- Phase 1
Brief Title: Pre-exposure Prophylaxis (PrEP) Rapid Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Victory Programs (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-43090
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Drug Use; Pre-exposure Prophylaxis (PrEP); Opioid Use Disorder
Keywords: People who inject drugs (PWID); Rapid PrEP Access; Substance use; Mobile health van
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Dried Blood Spot Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PrEP Rapid Access (Experimental): Participants who are at risk of HIV and being seen at the Victory Program's Mobile Prevention Services Van.
  Interventions: Other: PrEP Rapid Access; Other: HIV self-testing; Other: Dried blood spot testing

INTERVENTIONS:
Other: PrEP Rapid Access — 'Rapid PrEP Access' is a low-threshold intervention designed to provide on-site access to HIV self-testing at the Victory Program for persons who use opioids.
Other: HIV self-testing — After enrollment the research assistant (RA) will provide the participant with a HIV self-test and provide instructions on how to obtain a proper sample for the test. It uses an oral fluid test and yields results within 20 minutes.
Other: Dried blood spot testing — HIV Dried blood spot (DBS) testing provides an accurate method of measuring the HIV viral load in comparison to plasma viral load.

SUMMARY:
The goal of phase 1 is to determine the feasibility and acceptability of an intervention ('Rapid PrEP Access') providing people who use drugs (PWUD) one-time access to HIV self-testing at the Victory Program.

Aim 1: To offer HIV self-testing to PWUD in the community through a study called 'Rapid PrEP Access'. The study will be carried out at the Victory Program.

Aim 2: To determine the feasibility and acceptability of 'Rapid PrEP Access' at the Victory Program.

DETAILED DESCRIPTION:
For phase 1 of the study, participants will be recruited for a one-time baseline interview and HIV self-testing. A questionnaire will also be administered to assess their interest in the HIV prevention pill (PrEP= pre-exposure prophylaxis), but PrEP will not be offered. Study duration for each participant is one day; participants will not be followed over time.

After the prescreener and consent forms are completed, the Research Assistant (RA) will offer the participant an opportunity to administer an HIV self-test. The participant will be provided the test for unboxing and retrieving the user instructions.

All testing will be performed and interpreted by participants. The RA can provide assistance with reading the instruction on how to obtain a proper sample. Alternatively, the RA will direct them to information in the package insert which includes support offered by the OraQuick® Support Center.

After completing the HIVST, the RA will complete the baseline questionnaire with each participant while waiting for the participants' HIVST results. After the baseline questionnaire is complete, the RA will conduct satisfaction surveys to assess acceptability of the intervention and interest of PrEP initiation using REDCap.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Opioid use that was not prescribed by a health professional in the past 6 months

Exclusion Criteria:

* Pregnant women
* Persons with previous HIV diagnosis
* Individuals currently taking PrEP
* Individuals who express desire to harm themselves or others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Number of participants enrolled | 12 months
  Feasibility will be assessed by the number of participants enrolled
Acceptability of PrEP rapid Access | Through study completion, an average of 1 year
  Participants will rate PrEP Rapid Access' acceptability using an investigator-developed scale ranging from 1 to 5 where 1= not acceptable and 5 is very acceptable.

SECONDARY OUTCOMES:
Number of participants who perform HIV self-test | Through study completion, an average of 1 year
  This information will be obtained from information recorded on the day of recruitment for the study.
Number of participants interested in initiating PrEP | Through study completion, an average of 1 year
  This information will be obtained from information recorded on the day of recruitment from the survey data.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Assoumou, MD MPH, Principal Investigator — Boston Medical Center, Infectious Diseases
Locations (1):
- Victory Program, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Assoumou SA, Bonilla HV, Ruiz-Mercado G, Von Lossnitzer M, Baker R, Crawford ND, Bernstein JA. Community-based HIV Self-testing for Persons Who Use Drugs Can Contribute to Reaching Ending the HIV Epidemic in the US (EHE) Goals. Open Forum Infect Dis. 2024 Jun 17;11(6):ofae189. doi: 10.1093/ofid/ofae189. eCollection 2024 Jun. PMID 38887480